CLINICAL TRIAL: NCT02377570
Title: Comparison of the Clinical Performance of 3 THERANOVA 400 Dialyzer Prototypes With a High-Flux Dialyzer in Hemodialysis Mode - A Pilot Study
Brief Title: Comparison of the Clinical Performance of 3 THERANOVA 400 Dialyzer Prototypes With a High-Flux Dialyzer in Hemodialysis Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1407-003
Record Dates: First submitted 2015-02-10; First posted 2015-03-03 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- THERANOVA 400 dialyzer prototype AA (Experimental): THERANOVA 400 dialyzer prototype AA in hemodialysis treatment
  Interventions: Device: THERANOVA 400 dialyzer prototype AA
- THERANOVA 400 dialyzer prototype BB (Experimental): THERANOVA 400 dialyzer prototype BB in hemodialysis treatment
  Interventions: Device: THERANOVA 400 dialyzer prototype BB
- THERANOVA 400 dialyzer prototype CC (Experimental): THERANOVA 400 dialyzer prototype CC in hemodialysis treatment
  Interventions: Device: THERNOVA 400 dialyzer prototype CC
- FX CorDiax 80 dialyzer (Active Comparator): FX CorDiax 80 dialyzer in hemodialysis treatment
  Interventions: Device: FX CorDiax 80 dialyzer

INTERVENTIONS:
Device: THERANOVA 400 dialyzer prototype AA — Hemodialysis
  Arms: THERANOVA 400 dialyzer prototype AA
Device: THERANOVA 400 dialyzer prototype BB — Hemodialysis
  Arms: THERANOVA 400 dialyzer prototype BB
Device: THERNOVA 400 dialyzer prototype CC — Hemodialysis
  Arms: THERANOVA 400 dialyzer prototype CC
Device: FX CorDiax 80 dialyzer — Hemodialysis
  Arms: FX CorDiax 80 dialyzer

SUMMARY:
The study investigates the performance of a new dialyzer (Theranova 400) containing a membrane with increased pore sizes. The performance will be determined by the removal of middle molecules (with different molecular size) from the blood compartment. Three different Theranova 400 prototypes (AA, BB and CC) operated in hemodialysis mode will be compared with a Cordiax FX-80 dialyzer, operated in hemodialysis mode. Safety events and albumin loss into the dialysate will be monitored

ELIGIBILITY:
Inclusion Criteria:

1. Patient has end-stage renal disease
2. Patient is 18 years of age or older
3. Patient is male or female
4. Patient, if female, is non-pregnant; and if capable of becoming pregnant, will be using a medically acceptable means of contraception during participation in the study (Note: Female capable of becoming pregnant [defined as a woman less than 55 years old who has not had partial or full hysterectomy or oophorectomy] must have a negative serum beta human chorionic gonadotropin [β-hCG] test within 2 weeks of first study treatment)
5. Patient has been receiving HD or HDF therapy (HDF patients are allowed if their treatments during the study can be safely and effectively performed with HD) for ≥3 months prior to study enrollment and is expected to survive for at least 12 months after enrollment
6. Patient has a stable functioning native fistula, Gore-Tex graft, or double-lumen central venous catheter capable of providing a blood flow rate of ≥280 mL/min (with an acceptable recirculation rate, such that solute removal is not likely to be affected) based on the judgment of the treating physician
7. Patient is in clinically stable condition as judged by the treating physician and as demonstrated by stable medical history for 30 days prior to enrollment, physical examination, and laboratory testing
8. Patient is willing to comply with the study requirements for therapy during the entire study treatment period
9. Patient is capable of providing written informed consent to participate in the study

Exclusion Criteria:

1. Patient is undergoing single-needle dialysis
2. Patient has an abnormal κ/λ ratio (less than 0.37, or greater than 3.1)
3. Patient has a known active infection and is currently receiving antibiotic treatment
4. Patient has known active cancer
5. Patient has a known positive serology test for human immunodeficiency virus (HIV) or hepatitis B, C or E
6. Patient has a known serious hemostasis disorder
7. Patient has a known monoclonal gammopathy (eg, monoclonal gammopathy of uncertain significance, smouldering [asymptomatic] multiple myeloma, symptomatic multiple myeloma, nonsecretory multiple myeloma, plasmacytomas, or plasma cell leukemia)
8. Patient has a known polyclonal gammopathy (eg, connective tissue disease, liver disease, chronic infection, lymphoproliferative disorder, or other hematologic condition)
9. Patient has any other known comorbidity that could, in the opinion of the Investigator, potentially conflict with the study purpose or procedures (eg, severe hypoalbuminemia or anemia)
10. Patient has a known significant psychiatric disorder or mental disability that could interfere with the patient's ability to provide informed consent and/or comply with protocol procedures
11. Patient has a history of non-compliance with the dialysis prescription, as assessed by the Investigator
12. Patient has participated in another interventional clinical study in the past 3 months, or is currently participating in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall clearance of lambda immunoglobulin free light chains (molecular weight 45 kDa) | One mid-week dialysis session
  The primary efficacy endpoint is the overall clearance of lambda immunoglobulin free light chains during a mid-week hemodialysis session, assessed once with each experimental and active comparator product

SECONDARY OUTCOMES:
Instantanous clearance of a set of molecules with molecular sizes between 60 Da and 45 kDa | At 30 min from start of a mid-week dialysis session
  One secondary efficacy endpoint is the instantaneous clearance of a set of molecules with molecular sizes from 60 Da to 45 kDa at 30 min after start of a mid-week hemodialysis session, assessed once with each experimental and active comparator product
Instantanous clearance of a set of molecules with molecular sizes between 60 Da and 45 kDa | at 120 min from start of a mid-week dialysis session
  One secondary efficacy endpoint is the instantaneous clearance of a set of molecules with molecular sizes from 60 Da to 45 kDa at 120 min after start of a mid-week hemodialysis session, assessed once with each experimental and active comparator product
Overall clearance of a set of molecules with molecular sizes between 60 Da and 40 kDa | One mid-week dialysis session
  One secondary efficacy endpoint is the overall clearance of a set of molecules from 60 Da to 40 kDa during one mid-week hemodialysis session, assessed once with each experimental and active comparator product
Total mass removed of a set of molecules with molecular sizes between 60 Da and 45 kDa | One mid-week dialysis session
  One secondary efficacy endpoint is the total mass removed of a set of molecules from 60 Da to 45 kDa during one mid-week hemodialysis session, assessed once with each experimental and active comparator product
Removal rate of a set of molecules with molecular sizes between 60 Da and 45 kDa | One mid-week dialysis session
  One secondary efficacy endpoint is the removal rate of a set of molecules from 60 Da to 45 kDa during one mid-week hemodialysis session, assessed once with each experimental and active comparator product
Total mass removed of albumin | One mid-week dialysis session
  One secondary safety endpoint is the total removed mass of albumin during one mid-week hemodialysis session, assessed once with each experimental and active comparator product
Post- to pre-dialysis changes in a set of hematology parameters (blood cell counts, hematocrit and hemoglobin) | One mid-week dialysis session
  One secondary safety endpoint is the change in hematology parameters during one mid-week hemodialysis session, assessed once with each experimental and active comparator product
Types and frequency of adverse events and device deficiencies as a measure of safety and dialyzer tolerability | Continuously, from signature of informed consent form until 1 week after last hemodialysis session with an experimental or active comparator product, an expected average of 29 days
  Any adverse events and device deficiencies will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Haug, Manager, Study Director — Life Sciences & Operations, Gambro Dialysatoren GmbH ( a subsidiary of Baxter International Inc.)
Locations (1):
- LKH-Universität Klinikum Graz, Abteilung für Innere Medizin, Klinische Abteilung für Nephrologie und Dialyse, Graz, Austria

REFERENCES:
- [Result] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605
- [Result] Kirsch AH, Rosenkranz AR, Lyko R, Krieter DH. Effects of Hemodialysis Therapy Using Dialyzers with Medium Cut-Off Membranes on Middle Molecules. Contrib Nephrol. 2017;191:158-167. doi: 10.1159/000479264. Epub 2017 Sep 14. PMID 28910799